CLINICAL TRIAL: NCT01830400
Title: An Open-label, Multi-centre, Multi-national Post-marketing Non-interventional Prospective Study Evaluating Retention Rate, Seizure Control and Tolerability of Eslicarbazepine Acetate (ESL) as Adjunctive Treatment to One Baseline Antiepileptic Drug in Adult Patients With Partial-Onset Seizures With or Without Secondary Generalisation
Brief Title: A Post-marketing Study Evaluating Eslicarbazepine Acetate (ESL) as Adjunctive Treatment in Partial-Onset Seizures (Study E2093-E044-404) (EPOS)
Status: Completed | Type: Observational
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E2093-E044-404
Record Dates: First submitted 2013-04-08; First posted 2013-04-12 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Partial Onset Seizures
Keywords: ESL; Partial onset seizures; Retention Rate; Seizure Control; Antiepileptic; Secondary Generalisation
MeSH Terms: interventions — eslicarbazepine acetate

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Eslicarbazepine Acetate tablets
  Interventions: Drug: Eslicarbazepine Acetate tablets

INTERVENTIONS:
Drug: Eslicarbazepine Acetate tablets — The Eslicarbazepine Acetate (ESL) Summary of Product Characteristics (SPC) recommended a starting dose of 400 mg once-daily (QD) which was increased to 800 mg QD after one or two weeks. Based on individual response, the dose was increased to 1200 mg QD. Treatment decisions were made by clinicians in agreement with the participant, and were independent of participation in the study.
  Other Names: ESL

SUMMARY:
This was a Non-interventional Prospective Study. Centres enrolled adult patients with partial-onset seizures with or without secondary generalisation for whom the clinician had decided to initiate Eslicarbazepine Acetate (ESL) as an adjunctive therapy prior to the decision to take part in this study. Patients enrolled into the study were not sufficiently controlled with one drug licensed for the use as monotherapy in partial-onset seizures. Patients were seen at baseline and then during normal clinical visits at intervals. Patients in this study were assessed for efficacy and tolerability at baseline and then at least 3 and 6 months after the baseline.

ELIGIBILITY:
Inclusion Criteria:

* The decision to prescribe ESL was made by the physician before and independently of his/her decision to include the patient in the study
* Patients treated with one drug licensed for monotherapy in partial onset seizures
* Based on the physician's clinical judgment, the patient seizure activity was not controlled sufficiently with a current monotherapy and it was in the patient's best interest to be prescribed adjunctive ESL
* Patient was prescribed ESL no longer than 2 weeks before the baseline
* Treatment with ESL was to be commenced in line with the drug's license and Eslicarbazepine Acetate (ESL) Summary of Product Characteristics (SPC)
* Aged 18 years or older
* Signed written informed consent

Exclusion Criteria:

* Patients that had started ESL outside the approved SPC at enrolment
* Simultaneous participation in an interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Normal clinical practice setting/ centre.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Retention Rate of Eslicarbazepine Acetate (ESL) After 6 months from Baseline | 6 months

SECONDARY OUTCOMES:
Change in Overall Seizure Frequency after 3 and 6 months from Baseline | Baseline, 3 months and 6 months
  Change in overall seizure frequency calculated as absolute and percent changes after 3 and 6 months from baseline compared to the seizure frequency 3 months before introduction of ESL.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Holtkamp, Dr., Principal Investigator — Klinische und Experimentelle Epileptologie
Locations (106):
- Czechia (3):
  - Hradec Králové
  - Kroměříž
  - Prague
- Denmark (10):
  - Aalborg
  - Arhus C
  - Copenhagen
  - Dianalund
  - Esbjerg
  - Glostrup Municipality
  - Holstebro
  - Roskilde
  - Sønderborg
  - Vejle
- France (14):
  - Altkirch
  - Armentières
  - Bergerac
  - Biarritz
  - Chaumont
  - Cholet
  - Gap
  - Nice
  - Nîmes
  - Paris
  - Perpignan
  - Rueil-Malmaison
  - Sarreguemines
  - Toulon
- Germany (57):
  - Altenholz
  - Asperg
  - Augsburg
  - Bad Berka
  - Bad Langensalza
  - Berlin
  - Beuel
  - Bielefeld
  - Bochum
  - Bockhorn
  - Buxtehude
  - Cologne
  - Dortmund
  - Erbach im Odenwald
  - Erlangen
  - Etville
  - Gelsenkirchen
  - Gera
  - Greiz
  - Grevenbroich
  - Guelders
  - Hamburg
  - Hamm
  - Heilbad Heiligenstadt
  - Herdecke
  - Hildesheim
  - Hof
  - Ilmenau
  - Itzehoe
  - Kamp-Lintfort
  - Kirchen (Sieg)
  - Königsbrück
  - Leipzig
  - Leverkusen
  - Lohr a. Main
  - Ludwigsburg
  - Mannheim
  - Mittweida
  - München
  - Oranienburg
  - Osnabrück
  - Quakenbrück
  - Rathenow
  - Salzgitter
  - Schirgiswalde-Kirschau
  - Schorndorf
  - Schwäbisch Gmünd
  - Senftenberg
  - Solingen
  - Stuttgart
  - Troisdorf (Sieglar)
  - Waiblingen
  - Wesel
  - Westerstede
  - Wilhelmshaven
  - Wolfsburg
  - Würzburg
- Ireland (2):
  - Dooradoyle/ Co. Limerick
  - Dublin
- Norway (4):
  - Bergen
  - Molde
  - Oslo
  - Skien
- Sweden (5):
  - Angered
  - Helsingborg
  - Kungsbacka
  - Linköping
  - Stockholm / Saint Goran
- United Kingdom (11):
  - Birmingham
  - Dundee
  - London
  - Middlesbrough
  - Newport
  - Romford
  - Salford
  - Stoke-on-Trent
  - Telford
  - Torquay, Devon
  - Truro